CLINICAL TRIAL: NCT02026713
Title: "Impact of Cigarette Smoking on Platelet Reactivity in Patients With Acute Coronary Syndromes on Dual Antiplatelet Therapy With P2Y12 Inhibitors" - Trial COPTER -
Brief Title: Potential Impact of Cigarette Smoking on Platelet Reactivity in Patients on Dual Antiplatelet Therapy With P2Y12 Inhibitors
Acronym: COPTER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Polacco Marina, MD, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: WD-131213
Record Dates: First submitted 2013-12-18; First posted 2014-01-03 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- smokers on dual antiplatelet therapy with ASA and Prasugrel or (Experimental): All patients quit smoking for a 2 weeks period
  Interventions: Other: quit smoking for a 2 weeks period
- smokers on dual antiplatelet therapy with ASA and ticagrelor (Experimental): All patients on chronic dual antiplatelet therapy (>1 month) quit smoking for a 2 weeks period
  Interventions: Other: quit smoking for a 2 weeks period
- smokers on dual antiplatelet therapy with ASA and Clopidogrel (Active Comparator): All patients on chronic dual antiplatelet therapy (>1 month) quit smoking for a 2 weeks period
  Interventions: Other: quit smoking for a 2 weeks period

INTERVENTIONS:
Other: quit smoking for a 2 weeks period — evaluate the platelet reactivity after 15 days by quit smoking

SUMMARY:
All consecutive patients undergone PTCA in the period between July 2013 and December 2013 are eligible to be enrolled. Study population are divided in :

Group 1: smokers on dual antiplatelet therapy with ASA (100 mg once a day) and Prasugrel (10 mg die); Group 2: smokers on dual antiplatelet therapy with ASA(100 mg once a day) and Ticagrelor (90 mg twice a day); Control group: smokers on dual antiplatelet therapy with ASA(100 mg once a day) and Clopidogrel (75 mg once a day).

Platelet function is evaluated using a validated method: the VerifyNow System (Accumetrics Inc., San Diego, CA), which is a point-of-care turbidimetry-based optical detection system that measures platelet-induced aggregation. These value are measured Platelet function, measured with the VerifyNow P2Y12. All patients on chronic dual antiplatelet therapy (>1 month) quit smoking for a 2 weeks period. Therefore PRU values are obtained at baseline (at the enrollment time) and after 2 weeks after smoking cessation. Platelet reactivity are expressed in P2Y12 reaction units (PRU). PRU values >240 are suggestive of high platelet reactivity.

Primary outcomes: P2Y12 reaction units (PRU) at baseline and two weeks after quitting smoking.

DETAILED DESCRIPTION:
All consecutive patients undergone PTCA in the period between July 2013 and December 2013 are eligible to be enrolled. Study population are divided in :

Group 1: smokers on dual antiplatelet therapy with ASA (100 mg once a day) and Prasugrel (10 mg die); Group 2: smokers on dual antiplatelet therapy with ASA(100 mg once a day) and Ticagrelor (90 mg twice a day); Control group: smokers on dual antiplatelet therapy with ASA(100 mg once a day) and Clopidogrel (75 mg once a day).

Platelet function is evaluated using a validated method: the VerifyNow System (Accumetrics Inc., San Diego, CA), which is a point-of-care turbidimetry-based optical detection system that measures platelet-induced aggregation. These value are measured Platelet function, measured with the VerifyNow P2Y12. All patients on chronic dual antiplatelet therapy (>1 month) quit smoking for a 2 weeks period. Therefore PRU values are obtained at baseline (at the enrollment time) and after 2 weeks after smoking cessation. Platelet reactivity are expressed in P2Y12 reaction units (PRU). PRU values >240 are suggestive of high platelet reactivity.

Primary outcomes: P2Y12 reaction units (PRU) at baseline and two weeks after quitting smoking.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergone PTCA in our institution in the period between July 2013 and December 2013 will be eligible to be enrolled.
* smokers will be all patients smoking 15±10 cigarettes daily.
* patients on dual antiplatelet therapy with ASA and P2Y12 inhibitors.
* recent (<12 months) percutaneous coronary interventions
* angiographically-proven coronary artery disease

Exclusion Criteria:

- people unable to understand and willing to sign the informed consent form

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of platelet reaction units (PRU) | after 2 weeks of quitting smoking
  Absolute changes in platelet reactivity (expressed as P2Y(12) reaction units by the point-of-care VerifyNow assay [Accumetrics, San Diego, California])

CONTACTS AND LOCATIONS:
Overall Officials: marina MD polacco, medicine, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome, Rome, Roma, Italy

REFERENCES:
- [Derived] Patti G, Polacco M, Taurino E, Gaudio C, Greco C. Effects of cigarette smoking on platelet reactivity during P2Y12 inhibition in patients with myocardial infarction undergoing drug-eluting stent implantation: results from the prospective cigarette smoking on platelet reactivity (COPTER) study. J Thromb Thrombolysis. 2016 May;41(4):648-53. doi: 10.1007/s11239-016-1341-8. PMID 26849144